CLINICAL TRIAL: NCT03770728
Title: A 30-week, Multicenter, Double-blind, Placebo-controlled, Randomized Study to Evaluate the Efficacy and Safety of Efpeglenatide Once Weekly in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin Alone or in Combination With Sulfonylurea
Brief Title: Efficacy and Safety of Efpeglenatide Versus Placebo in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin Alone or in Combination With Sulfonylurea
Acronym: AMPLITUDE-S
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to cancel TRIAL, not related to safety concern
Sponsor: Sanofi (Industry)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15337; U1111-1205-1291 (Other: UTN)
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo (matched to Efpeglenatide) subcutaneous (SC) injection once weekly up to Week 30 on top of metformin alone or in combination with SU.
  Interventions: Drug: Placebo; Drug: Background therapy: Metformin alone or in combination with SU
- Efpeglenatide 2 mg (Experimental): Participants received Efpeglenatide 2 milligrams (mg) SC injection once weekly up to Week 30 on top of metformin alone or in combination with SU.
  Interventions: Drug: Efpeglenatide SAR439977; Drug: Background therapy: Metformin alone or in combination with SU
- Efpeglenatide 4 mg (Experimental): Participants received Efpeglenatide 4 mg SC injection once weekly up to Week 30 on top of metformin alone or in combination with SU. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg and was maintained at the 4 mg dose through-out the treatment duration, up to Week 30.
  Interventions: Drug: Efpeglenatide SAR439977; Drug: Background therapy: Metformin alone or in combination with SU
- Efpeglenatide 6 mg (Experimental): Participants received Efpeglenatide 6 mg SC injection once weekly up to Week 30 on top of metformin alone or in combination with SU. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg until Week 3 and later up-titrated to 6 mg and was maintained at the 6 mg dose through-out the treatment duration, up to Week 30.
  Interventions: Drug: Efpeglenatide SAR439977; Drug: Background therapy: Metformin alone or in combination with SU

INTERVENTIONS:
Drug: Efpeglenatide SAR439977 — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Efpeglenatide 2 mg; Efpeglenatide 4 mg; Efpeglenatide 6 mg
Drug: Placebo — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Placebo
Drug: Background therapy: Metformin alone or in combination with SU — Pharmaceutical form: tablet Route of administration: oral, administered as per investigator and in accordance with local labeling.

SUMMARY:
Primary Objective:

To demonstrate the superiority of once weekly injection of efpeglenatide in comparison to placebo in glycated hemoglobin (HbA1c) change in participants with type 2 diabetes mellitus (T2DM) inadequately controlled with metformin alone or in combination with sulfonylurea (SU).

Secondary Objectives:

* To demonstrate the superiority of once weekly injection of efpeglenatide in comparison to placebo on glycemic control.
* To demonstrate the superiority of once weekly injection of efpeglenatide in comparison to placebo on body weight.
* To evaluate the safety of once weekly injection of efpeglenatide.

DETAILED DESCRIPTION:
Study duration per participant was approximately 39 weeks including an up to 3-week Screening Period, a 30-week Treatment Period, and a 6-week safety Follow-up Period.

ELIGIBILITY:
Inclusion criteria:

* Participant must be greater than or equal to (>=)18 years of age at the time of signing the informed consent.
* Participants with T2DM.
* Diabetes diagnosed at least 1 year before screening.
* Participants on metformin alone or in combination with SU, for at least 3 months prior to screening.
* Glycated hemoglobin between 7.0% and 10.0% (inclusive) measured by the central laboratory at screening.

Exclusion criteria:

* History of severe hypoglycemia requiring emergency room admission or hospitalization within 3 months prior to screening.
* Retinopathy or maculopathy with one of the following treatments, either recent (within 3 months prior to screening) or planned: intravitreal injections or laser or vitrectomy surgery.
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to) gastroparesis, unstable and not controlled gastroesophageal reflux disease requiring medical treatment within 6 months prior to screening or history of surgery affecting gastric emptying.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy.
* Personal or family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (e.g., multiple endocrine neoplasia syndromes).
* Body weight change of >=5 kilograms within the last 3 months prior to screening.
* Systolic blood pressure greater than (>)180 millimeters of mercury (mmHg) and/or diastolic blood pressure >100 mmHg at randomization.
* Severe renal disease as defined by estimated glomerular filtration rate (eGFR) of <30 milliliters per minute per 1.73 square meter.
* Laboratory findings at the screening visit:

  * Alanine aminotransferase or aspartate aminotransferase >3*upper limit of the normal (ULN) or total bilirubin >1.5*ULN (except in case of documented Gilbert's syndrome);
  * Amylase and/or lipase: >3*ULN laboratory range;
  * Calcitonin >=5.9 picomoles per liter (20 picograms per milliliter).
* Gastric surgery or other gastric procedures intended for weight loss within 2 years prior to screening, or planned during study period.
* Pregnant (confirmed by serum pregnancy test at screening) or breast-feeding women.
* Women of childbearing potential not willing to use highly effective method(s) of birth control or who are unwilling to be tested for pregnancy during the study period and for at least 5 weeks after the last dose of study intervention.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (48):
- United States (23):
  - Investigational Site Number 8400038, Birmingham, Alabama
  - Investigational Site Number 8400035, Chandler, Arizona
  - Investigational Site Number 8400005, Glendale, Arizona
  - Investigational Site Number 8400042, Mesa, Arizona
  - Investigational Site Number 8400051, Phoenix, Arizona
  - Investigational Site Number 8400056, Tucson, Arizona
  - Investigational Site Number 8400057, Huntington Park, California
  - Investigational Site Number 8400009, Los Angeles, California
  - Investigational Site Number 8400045, Spring Valley, California
  - Investigational Site Number 8400040, Tustin, California
  - Investigational Site Number 8400047, Colorado Springs, Colorado
  - Investigational Site Number 8400046, Coral Gables, Florida
  - Investigational Site Number 8400041, Pembroke Pines, Florida
  - Investigational Site Number 8400025, Lawrenceville, Georgia
  - Investigational Site Number 8400044, Lexington, Kentucky
  - Investigational Site Number 8400001, Bridgeton, New Jersey
  - Investigational Site Number 8400039, New Windsor, New York
  - Investigational Site Number 8400036, Morehead City, North Carolina
  - Investigational Site Number 8400013, Maumee, Ohio
  - Investigational Site Number 8400048, Oklahoma City, Oklahoma
  - Investigational Site Number 8400030, Dallas, Texas
  - Investigational Site Number 8400043, San Antonio, Texas
  - Investigational Site Number 8400037, Layton, Utah
- China (22):
  - Investigational Site Number 1560005, Baotou
  - Investigational Site Number 1560042, Beijing
  - Investigational Site Number 1560053, Hangzhou
  - Investigational Site Number 1560051, Hefei
  - Investigational Site Number 1560011, Hunan
  - Investigational Site Number 1560025, Meihekou
  - Investigational Site Number 1560055, Nanchang
  - Investigational Site Number 1560024, Nanjing
  - Investigational Site Number 1560020, Pingxiang
  - Investigational Site Number 1560031, Shandong
  - Investigational Site Number 1560030, Shandong
  - Investigational Site Number 1560012, Shanghai
  - Investigational Site Number 1560013, Shanghai
  - Investigational Site Number 1560004, Shanghai
  - Investigational Site Number 1560022, Shanghai
  - Investigational Site Number 1560041, Tianjin
  - Investigational Site Number 1560010, Wenzhou
  - Investigational Site Number 1560052, Wuhu
  - Investigational Site Number 1560034, Wuxi
  - Investigational Site Number 1560026, Xuzhou
  - Investigational Site Number 1560044, Yichun
  - Investigational Site Number 1560003, Zhengzhou
- Taiwan (3):
  - Investigational Site Number 1580006, Kaohsiung City
  - Investigational Site Number 1580003, Taichung
  - Investigational Site Number 1580002, Taipei

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) by SANOFI: Product rights transferred to Hanmi Pharmaceutical.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 48 active sites in 3 countries. A total of 560 participants were screened between 01 August 2019 and 09 August 2020, out of which 248 were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: A total of 312 participants were randomized in 1:1:1:1 ratio to either placebo, efpeglenatide 2 milligrams (mg), efpeglenatide 4 mg, or efpeglenatide 6 mg treatment arms, stratified by screening glycated hemoglobin (HbA1c) values (less than [<]8%, greater than or equal to [>=]8%) and sulfonylurea (SU) use at screening (Yes/No).
Groups:
- Efpeglenatide 2 mg: Participants received Efpeglenatide 2 mg SC injection once weekly up to Week 30 on top of metformin alone or in combination with SU.
Period: Overall Study
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Started | 79 | 78 | 77 | 78
Safety Population (Participants who received at least 1 dose or part of a dose of the Investigational Medicinal Product (IMP), analyzed according to the treatment actually received.) | 79 | 78 | 80 (For safety analysis, participants were included in the treatment group that they were exposed for longer duration. 3 participants randomized to Efpeglenatide 6 mg received 4 mg dose for longer duration; and considered in Efpeglenatide 4 mg group for safety analysis.) | 75
Completed | 41 | 47 | 45 | 43
Not Completed | 38 | 31 | 32 | 35
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Poor compliance to protocol | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 13 | 8 | 9 | 13
Not completed — Other than specified | 24 | 23 | 21 | 22

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-treat (ITT) population, which included all participants randomized irrespective of rescue therapy use and compliance with the study protocol and procedures, and were analyzed according to the treatment group allocated by randomization.
Groups:
- Placebo: Participants received placebo (matched to Efpeglenatide) SC injection once weekly up to Week 30 on top of metformin alone or in combination with SU.
- Total: Total of all reporting groups
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Total
Number analyzed (Participants) | 79 | 78 | 77 | 78 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.6) | 60.1 (10.9) | 57.9 (10.5) | 58.8 (11.5) | 58.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 33 | 39 | 140
  Male | 45 | 44 | 44 | 39 | 172
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 43 | 46 | 48 | 179
  Black or African American | 11 | 10 | 4 | 7 | 32
  Asian | 24 | 24 | 26 | 22 | 96
  Other | 2 | 1 | 1 | 0 | 4
  Not reported | 0 | 0 | 0 | 1 | 1
Baseline Glycated Hemoglobin (HbA1c %) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.09 (0.79) | 8.07 (0.76) | 8.15 (0.69) | 8.09 (0.79) | 8.10 (0.76)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 32.2 (7.1) | 31.8 (7.7) | 32.0 (6.3) | 32.4 (7.4) | 32.1 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 30 in HbA1c
Description: This analysis included all Week 30 assessment values available.
Time Frame: Baseline to Week 30
Population: Analysis was performed on Intent-to-treat (ITT) population, which included all participants randomized irrespective of rescue therapy use and compliance with the study protocol and procedures, and were analyzed according to the treatment group allocated by randomization. Here, "Overall number of participants analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 48 | 48 | 49 | 48
percentage of HbA1c | -0.27 (0.92) | -1.05 (0.88) | -1.46 (0.90) | -1.36 (1.09)

2. Secondary Outcome: Number of Participants With HbA1c <7.0%
Description: Participants who had no available assessment for HbA1c <7% at Week 30 were considered as non-responders.
Time Frame: Week 30
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 79 | 78 | 77 | 78
Participants | 11 | 27 | 33 | 32

3. Secondary Outcome: Change From Baseline to Week 30 in Fasting Plasma Glucose (FPG)
Description: This analysis included all Week 30 assessment values available.
Time Frame: Baseline to Week 30
Population: Analysis was performed on ITT population. Here, "Overall number of participants analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 45 | 45 | 47 | 43
millimoles per liter (mmol/L) | 0.12 (2.37) | -0.97 (2.43) | -1.75 (2.43) | -1.20 (4.68)

4. Secondary Outcome: Change From Baseline to Week 30 in Body Weight
Description: This analysis included all Week 30 assessment values available.
Time Frame: Baseline to Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 47 | 46 | 47 | 47
kilograms | -1.89 (5.53) | -2.49 (3.93) | -2.72 (6.49) | -3.87 (4.62)

5. Secondary Outcome: Number of Participants With At Least One Hypoglycemic Events (Documented Symptomatic Hypoglycemia <3.0 mmol/L [<54 mg/dL], Severe Hypoglycemia)
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <54 milligrams per deciliter (mg/dL) (<3.0 mmol/L). Severe hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Baseline up to Week 30
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Efpeglenatide 4 mg: Participants received Efpeglenatide 4 mg SC injection once weekly up to Week 30 on top of metformin alone or in combination with SU. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg and maintained at the 4 mg dose through-out the treatment duration, up to Week 30.
- Efpeglenatide 6 mg: Participants received Efpeglenatide 6 mg SC injection once weekly up to Week 30 on top of metformin alone or in combination with SU. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg until Week 3 and later up-titrated to 6 mg and maintained at the 6 mg dose through-out the treatment duration, up to Week 30.
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 79 | 78 | 80 | 75
Participants
  Documented symptomatic hypoglycemia (<54 mg/dL) | 1 | 0 | 2 | 3
  Severe hypoglycemia | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Hypoglycemic Events (Documented Symptomatic Hypoglycemia <3.0 mmol/L [<54 mg/dL] and Severe Hypoglycemia) Per Participant-Year
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <54 mg/dL (<3.0 mmol/L). Severe hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Baseline up to Week 30
Population: Analysis was performed on safety population.
Measure: Number; unit: events per participant-year
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 79 | 78 | 80 | 75
events per participant-year
  Documented symptomatic hypoglycemia (<54 mg/dL) | 0.03 | 0 | 0.06 | 0.14
  Severe hypoglycemia | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent up to end of study (up to Week 36). Time frame for reporting of treatment emergent adverse events (TEAEs) was from first injection of investigational medicinal product (IMP) up to 30 days after the last injection of the IMP (i.e. up to Week 34).
Description: TEAEs were defined as AEs that developed or worsened or became serious during the treatment-emergent period. Analysis was performed on safety population.
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/78 | 0/80 | 0/75
Serious Adverse Events (participants affected / at risk) | 3/79 | 4/78 | 5/80 | 2/75
Other Adverse Events (participants affected / at risk) | 21/79 | 30/78 | 36/80 | 32/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=79) | Efpeglenatide 2 mg (N=78) | Efpeglenatide 4 mg (N=80) | Efpeglenatide 6 mg (N=75)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=79) | Efpeglenatide 2 mg (N=78) | Efpeglenatide 4 mg (N=80) | Efpeglenatide 6 mg (N=75)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 1 (1) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (10) | 5 (5) | 2 (2) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 3 (3) | 6 (7) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4) | 4 (5)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (9) | 13 (16) | 12 (17)
Nausea (Gastrointestinal disorders) | 5 (6) | 10 (10) | 16 (17) | 8 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 6 (6) | 10 (16)
Fatigue (General disorders) | 1 (1) | 4 (5) | 5 (5) | 0 (0)
Injection Site Pain (General disorders) | 4 (5) | 2 (4) | 2 (2) | 2 (2)
Lipase Increased (Investigations) | 1 (2) | 4 (5) | 6 (7) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor on 09 September 2020. Due to early termination of the study, few efficacy evaluations and analyses originally planned in the protocol were no longer considered to be applicable and were not performed. Primary, and secondary efficacy data were descriptively summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03770728/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03770728/SAP_001.pdf